CLINICAL TRIAL: NCT07017023
Title: Cognitive Effects of Losartan-augmented Behavioural Activation in Anhedonia
Brief Title: Combined Blood Pressure Medication and Activity Scheduling for Low Mood
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CUREC reference 660982
Record Dates: First submitted 2025-05-19; First posted 2025-06-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Emotional Processing; Mood
Keywords: emotional processing; mood
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Parallel randomised experimental medicine trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan (Experimental): 7-day losartan potassium (Cozaar; 50mg; oral tablet) with 7-day BA
  Interventions: Drug: Losartan with BA
- Placebo (Placebo Comparator): 7-day placebo (oral; microcellulose in identical capsules) with 7-day BA
  Interventions: Other: Placebo with BA

INTERVENTIONS:
Drug: Losartan with BA — 7-day losartan (Cozaar, 50mg; oral tablet) with 7-day BA
  Arms: Losartan
Other: Placebo with BA — 7-day placebo (oral; microcellulose in identical capsules) with 7-day BA
  Arms: Placebo

SUMMARY:
This study explores the effects of 7-day losartan (50mg) versus placebo with brief behavioural activation on emotional processing in young volunteers low in positive mood

DETAILED DESCRIPTION:
Behavioural Activation (BA) is a first-line treatment for depression that aims to re-engage patients with rewarding activities, to improve mood. However, patients with low levels of positive mood respond less well to BA than others. Neuroscience has identified deficits in the processing of positive stimuli in this group of people, using cognitive-psychological computer tasks and brain imaging. Losartan, a licensed medication targeting the renin-angiotensin system, has recently been found to improve the processing of positive stimuli in healthy volunteers. Combining losartan with BA may improve treatment response in people with low positive mood, by improving positive information processing. This study will test this hypothesis.

In a double-blind randomised trial, 76 participants with low positive mood will receive 7-day behavioural activation (BA) with daily losartan (50mg) or placebo. Before and after the intervention, they will complete computer tasks measuring processing of positive and negative information.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Aged 18-65 years
* Self-reported low levels of positive mood
* Sufficient written and spoken English skills to understand study procedures
* Normal or corrected to normal vision and hearing
* Access to a computer and reliable internet connection

Exclusion Criteria:

* Antidepressant treatment or medication in last three months
* Currently receiving cognitive-behavioural therapy with behavioural activation
* History of psychosis or bipolar disorder
* History of substance dependence
* Use of illegal drugs in last 3 months
* First-degree relative with history of psychosis or bipolar disorder
* Current or past hospitalisation for mental health reasons
* BDI-II score >30
* Judged to be currently at clinical risk of suicide
* Past suicide attempt
* CNS-medication last 6 weeks (including in another study)
* Severely underweight or overweight in a manner that renders them unsuitable for the study in the opinion of the study medic
* Current blood pressure or other heart medication
* Diagnosis of intravascular fluid depletion or dehydration
* History of angioedema
* Impaired kidney function (based on self-report)
* Very low blood pressure following established definitions (at least three consecutive measurements of blood pressure under standardised conditions where either the systolic or the diastolic blood pressure or both are below 90/60 mmHg (in accordance with established standard definitions: https://www.nhs.uk/cond...-pressure-hypotension/)
* Current diagnosis of a developmental disorder (e.g. ADHD, Tourette's syndrome, severe learning disability) according to self-report, where in the opinion of the study team such difficulties would likely interfere with compliance or task performance
* Current diagnosis of a neurological disorder (e.g. epilepsy, MS) according to self-report
* Lifetime history of systemic infection, or clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, metabolic, endocrine or pulmonary disease or disorder which, in the opinion of the investigator, may put the participant at risk when participating, or may influence compliance or task performance
* Pregnancy (urine pregnancy test during Baseline Visit), breast feeding or plans to become pregnant during study participation
* Heavy use of cigarettes (smoke > 20 cigarettes per day)
* Severe lactose intolerance (due to losartan containing some lactose monohydrate)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in reinforcement learning | from baseline to post 7-day intervention
  reinforcement learning, calculated as the learning rate from negative and positive decision outcomes. Larger scores indicate better learning from an outcome.

SECONDARY OUTCOMES:
Change in approach-avoidance-task (AAT) effect score | from baseline to post 7-day intervention
  mean reaction time of the pull trials of a valence category subtracted from the push trials of the same category, yielding a single indicator of approach/avoidance, with positive scores indicating relatively stronger approach and negative scores indicating relatively stronger avoidance
Change in social approach decisions | from baseline to post 7-day intervention
  % approach vs avoid decisions
Change in motivational effort in the Apples Task | from baseline to post 7-day intervention
  The task weighs effort costs against reward value. It involves a hand dynamometer to record effort. On each trial, participants receive an offer showing a reward (number of apples shown on a tree) and an effort level (height of marking on the tree trunk), which they can accept or reject (Yes/No response). On a subset of accepted trials, participants have to exert physical effort on the hand dynamometer to earn the reward (number of apples in the respective trial). Participants receive monetary reward for the number of apples collected. Key outcome marker is effort-reward valuation, i.e. % accepted trials based on combinations of effort and reward levels. Other outcomes: Force exerted relative to Maximum Voluntary Contraction (MVC), Reaction times of Yes/No.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Reinecke, PhD, Principal Investigator — University of Oxford
Locations (1):
- Warneford Hospital, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided